CLINICAL TRIAL: NCT03413475
Title: Oral Quality of Life of Patients to be Totally Edentulous at One Arch at Least and Benefiting From the Realization of Immediate and Usual Complete Removable Prostheses.
Brief Title: Oral Quality of Life
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0260
Record Dates: First submitted 2018-01-15; First posted 2018-01-29 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Odontalgia
Keywords: Edentulism; complete removable prosthesis; quality of life
MeSH Terms: conditions — Toothache | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: quality of life

SUMMARY:
The restorative and surgical odontological department at the Nantes University Hospital frequently hosts patients with a severely degraded oral condition who has never benefited from a removable prosthetic rehabilitation. The chosen treatment plan consists most of the time in extracting all the residual teeth at one or both arches with the immediate insertion of a complete removable prosthesis performed prior to the extractions. This prosthesis is adapted by regular relining during the osteomucosal healing and is replaced by a usage removable prosthesis on average 6 months after the extractions.

The transition from dentate state (even dilapidated) to toothless state can be a source of discomfort and impairment and lead to a decrease of life's quality for patients. The purpose of this study is to evaluate oral health of the patients at the different stages of prosthetic rehabilitation by using GOHAI (Geriatric Oral Health Assessment Index).

DETAILED DESCRIPTION:
Patients are selected at the beginning of their prosthetic rehabilitation and selected patients give their consent for the participation at the clinical trial. The filling of the GOHAI questionnaire is performed in 3 steps:1- before treatment, 2- after teeth extractions and the delivering of immediate complete denture or without immediate prosthetic rehabilitation and 3-during inspection visits after the delivery of the definitive denture.

ELIGIBILITY:
Inclusion Criteria:

* An adult man or a woman, speaking and understanding French, benefiting from social security cover.
* Patient presenting one or more teeth to be extracted, these extractions resulting in a complete uni or bimaxillary edentulism rehabilitated or not by an immediate complete removable prosthesis.

Exclusion Criteria:

* Patients under the age of majority, patients under protection, protected persons, patients refusing to participate in the study, patients whose follow-up can't be performed, patients who don't speak French and patients who don't benefit from social coverage.
* Patients rehabilitated by immediate partial removable prosthesis (persistence of teeth on the rehabilitated arch).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated for prosthetic rehabilitation with the need for a total edentemant of at least one arch, and setting up a complete removable prosthesis
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Geriatric Oral Health Assessment Index (GOHAI) questionnaire | Day - 30
  GOHAI questionnaire (Geriatric Oral Health Assessment Index) (12 questions) before the treatment when the patient is still partially dentate (Day -30).
Geriatric Oral Health Assessment Index (GOHAI) questionnaire | Day 0
  GOHAI questionnaire (Geriatric Oral Health Assessment Index) (12 questions) in the control sessions after delivery of immediate prostheses (day 0)
Geriatric Oral Health Assessment Index (GOHAI) questionnaire | month 1
  OHAI questionnaire (Geriatric Oral Health Assessment Index) (12 questions) in the control sessions during the healing phase for patients not rehabilitated at 1 month,
Geriatric Oral Health Assessment Index (GOHAI) questionnaire | Month 3
  after carrying out the usage prostheses during the inspection visits at 3 months (with a patient carrying his prostheses for at least 1 month).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Le Guehennec, DDS, PhD, Principal Investigator — Nantes University Hospital
Locations (1):
- Hospital University of Nantes, Nantes, France